CLINICAL TRIAL: NCT05780697
Title: Short Term Results of Pediatric Septic Hip Arthritis Management in Assiut University Hospitals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Beshoy Elkess Ibram, Resident Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pediatric Septic Hip arthritis
Record Dates: First submitted 2023-03-13; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Septic Arthritis
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children presented with septic hip arthritis in Assiut University Hospitals (Experimental): Surgery of Drainage of pus in septic hip arthritis
  Interventions: Procedure: Surgery of Drainage of septic hip arthritis

INTERVENTIONS:
Procedure: Surgery of Drainage of septic hip arthritis — Surgery for septic hip arthritis by anterior or lateral approach and inspection of femoral head

SUMMARY:
Detect short term results of pediatric septic hip arthritis and its risk factors

DETAILED DESCRIPTION:
Septic arthritis of the hip is a true orthopedic emergency(1). In developed countries, the incidence of acute bacterial septic arthritis is estimated to be 4 to 10 per 100,000 children (2).It is caused by many microorganisms. Staph aureus is most common in children over 2 years of age . Staph aureus is gram-positive cocci in clusters and most common in nosocomial infections of neonates(3-4).Group B streptococcus is most common in neonates with community-acquired infection and exposed during transvaginal delivery(5).Neisseria gonorrhoeae is gram-negative diplococci and most common in adolescents.when the causative Organism is Neisseria gonorrhoeae ,patients usually have a preceding migratory polyarthralgia,multiple joint involvement and small red papules(6-7).Group A beta-hemolytic streptococcus is most common organism following varicella infection.HACEK organisms (Haeophilus,Actinobacillus,Cardiobacterium,Eikenella,and Kingella fastidious) are less common causative organisms(8-9).Early diagnosis and accurate treatment is key in avoiding complications such as joint destruction,joint dislocation , ankylosis, growth arrest or spread of infection leading to osteomyelitis , pelvic abscess or nerve lesions.. Treatment is started without delay after synovial fluid and blood samples have been obtained. The classical presentation of septic hip arthritis in children is a combination of a painful hip joint with limited range of motion, fever, malaise and inability to bear weight on the affected limb. Misdiagnosis or inappropriate treatment of acute septic arthritis of the hip in children can result in devastating damage of the joint and possible lifelong disability. Open arthrotomy , drainage and thorough irrigation of the joint is considered the standard treatment for septic arthritis of the hip.Empiric antibiotic treatment primarily targets S. aureus and takes into account its resistance to antibiotics(10-11). So,we want to detect short term results of pediatric septic hip arthritis at Assiut University Hospitals

ELIGIBILITY:
Inclusion Criteria:

- Children younger than 14 years old presented with septic hip arthritis only or by bilateral septic hip arthritis in Assiut University Hospitals

Exclusion Criteria:

* 1-patients with Tuberculous arthritis 2-patients whose parents refuse to participate in the study

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Modified Moon's criteria for outcome assessment of hip function | Baseline

SECONDARY OUTCOMES:
Detection of Complications | Baseline
  Complications such as limb-lenght discrepancy , Avascular necrosis of the femoral head and hip destruction will be documented

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fabry G, Meire E. Septic arthritis of the hip in children: poor results after late and inadequate treatment. J Pediatr Orthop. 1983 Sep;3(4):461-6. doi: 10.1097/01241398-198309000-00008. PMID 6630490
- [Background] Ilharreborde B. Sequelae of pediatric osteoarticular infection. Orthop Traumatol Surg Res. 2015 Feb;101(1 Suppl):S129-37. doi: 10.1016/j.otsr.2014.07.029. Epub 2014 Dec 29. PMID 25553604